CLINICAL TRIAL: NCT01798173
Title: CIRCE: Environmental, Metabolic and Nutritional Factors of Hepatocellular Carcinoma in Cirrhotic Patients
Brief Title: Environmental, Metabolic and Nutritional Factors of Hepatocellular Carcinoma in Cirrhotic Patients
Acronym: CIRCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HILLON HORS AOI 2008
Record Dates: First submitted 2013-01-04; First posted 2013-02-25 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Cirrhosis With Hepatocellular Carcinoma; Cirrhosis Without Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Cirrhosis; Environmental risk factors; Nutrition; Metabolic syndrome
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis; Metabolic Syndrome | interventions — Magnetic Resonance Spectroscopy

ARMS (2):
- Cases: cirrhotic patients with hepatocellular carcinoma (Experimental)
  Interventions: Biological: Serum, plasma and DNA samples; Procedure: Radiological exploration by CT scan or MRI
- Controls: cirrhotic patients without hepatocellular carcinoma (Active Comparator)
  Interventions: Biological: Serum, plasma and DNA samples; Procedure: Radiological exploration by CT scan or MRI

INTERVENTIONS:
Biological: Serum, plasma and DNA samples
Procedure: Radiological exploration by CT scan or MRI

SUMMARY:
Available data do not allow carcinogenesis mechanisms in cirrhotic patients to be well understood in absence of studies taking into account all recognised factors. A large scale clinical, biochemical and molecular studies is potentially relevant to the understanding of nutrition, physical activity, body weight metabolic syndrome whatever the etiology of underlying cirrhosis. It will open new perspectives :

* in prevention of hepatocellular carcinoma development in cirrhotic patients through dietary counselling and therapeutics of metabolic syndrome,
* in early screening of hepatocellular carcinoma in cirrhotic patients through spectroscopic technology and later proteomic study resulting in an improvement of hepatocellular carcinoma prognosis.

ELIGIBILITY:
Inclusion Criteria:

Cases and controls will be males and females aged 35 or older, and will give an informed consent to participate in the study.

* Hepatocellular carcinoma case:

All hepatocellular carcinoma cases evolving in cirrhotic liver, whatever the etiology of cirrhosis, will be included. Criteria for the diagnosis of hepatocellular carcinoma will be those defined by the European Association for Study of the Liver (EASL) (Bruix J, J Hepatol 2001):

Focal hepatic lesions ≥ 2cm in diameter:

* alpha-fetoprotein (AFP) < 400 ng/ml: nodules have to be identified by at least two coincident morphologic examinations (abdominal US, angiography, CT or MRI) with arterial hypervascularisation in at least one of the imaging modalities
* AFP > 400 ng/ml: lesion seen in a single imaging modality

Focal hepatic lesions < 2 cm in diameter:

* lesions 1 to 2 cm in diameter:use of fine-needle aspiration with biopsy
* lesions < 1 cm: serial abdominal US every 3 months until the lesion exceeds 1 cm in size so that biopsy becomes possible. Such cases will be included after diagnosis confirmation.

Whatever the size of focal lesions, the diagnosis of cirrhosis will be made according to the same criteria as in the cirrhotic group control.

* Cirrhotic control patients:

All patients with cirrhosis, whatever its etiology, will be included. The diagnosis of cirrhosis will rely on:

Histological confirmation by liver biopsy or in the absence of biopsy:

* in patients free of portal thrombosis at Doppler imaging, on the presence of portal hypertension ascertained by biological (tricytopenia), morphologic (abdominal US, CT or MRI), hepatic venous pressure measurement or upper endoscopy (mosaic gastropathy, varices).
* in patients with portal thrombosis, on the presence of portal hypertension associated with: Clinical (hepatomegaly with clinical evidence of hepatocellular failure: spider naevi, palmar erythema, white mails, gynecomastia) or morphological signs of cirrhosis (enlarged liver, nodular surface, sharp lower edge).

And/or biological signs of hepatocellular failure (TP<70%, low albuminemia) And/or sinusoidal block assessed by liver venous gradient > 18mmHG In the present state of knowledge, a fibrotest value at 4 or a fibroscan value > 12.5 kilopascal.

Without any other clinical or biological signs will be considered as diagnosis criteria of cirrhosis only for chronic viral C hepatitis.

The lack of hepatocellular carcinoma in cirrhotic patients at inclusion will be assessed through good quality imaging examinations (abdominal US, CT scan or MRI) and AFP below 100 ng/ml.

Exclusion Criteria:

* age under 35 of year
* other cancer in evolution
* HIV infection
* Major somatic pr psychiatric illness not compatible with the inclusion in the study
* No hepatocellular carcinoma primary liver cancer.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1246 (Actual)
Dates: Start 2008-06-20 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25

PRIMARY OUTCOMES:
Dosage of the vitamin B12 and the folates | Baseline

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Hôpital Jean Minjoz, Besançon
  - Hôpital du Bocage, Dijon
  - Centre Hospitalier de METZ, Metz
  - CHU Robert DEBRE, Reims
  - Clinique médicale B. Hôpital Civil-Hôpitaux Universitaires, Strasbourg
  - Hôpital de BRABOIS, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Rizk M, Roux-Levy C, Bernard-Chabert B, Bronowicki JP, Richou C, Habersetzer F, Jouve JL, Hebert JR, Shivappa N, Boutron-Ruault MC, Diab Assaf M, Hillon P, Cottet V; other members of the CirCE Study group. Association between the dietary inflammatory index and the risk of hepatocellular carcinoma in a cirrhotic population. Clin Nutr. 2025 Jan;44:65-75. doi: 10.1016/j.clnu.2024.11.021. Epub 2024 Nov 14. PMID 39642746